CLINICAL TRIAL: NCT03787953
Title: A Real World Study of Anti-PD-1/PD-L1 Antibodies for the Treatment of Advanced Solid Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Xiao Zhao, Principal Investigator, Chinese PLA General Hospital
Other Study IDs: PDL1-2018-301BJ
Record Dates: First submitted 2018-12-20; First posted 2018-12-27 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Advanced Solid Tumors
Keywords: anti-PD-1/PD-L1 antibodies; Efficacy; Safety; Real world study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Biopsy specimen or blood specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anti-PD-1/PD-L1 antibodies: Patients with advanced solid tumors who visited Department of Medical Oncology, Chinese PLA General Hospital from 2015 to 2019 and received anti-PD-1/PD-L1 antibody therapy
  Interventions: Drug: Anti-PD-1/PD-L1 antibodies

INTERVENTIONS:
Drug: Anti-PD-1/PD-L1 antibodies — The study is a real-world study. According to the actual medical history of patients, the usage of anti-PD-1/PD-L1 antibodies was collected.

SUMMARY:
The study was designed to analyze the efficacy and safety of anti-PD-1/PD-L1 antibodies for the treatment of advanced solid tumors.

DETAILED DESCRIPTION:
The study is a real-world study and the case records of patients with advanced solid tumors who visited Department of Medical Oncology, Chinese PLA General Hospital from 2015 to 2019 and received anti-PD-1/PD-L1 antibody therapy will be collected in this study. The medical data including patient demographic, tumor characteristics, laboratory examination, history of treatments, adverse reactions, and so on will be extracted to analyze the effectivity and safety of anti-PD-1/PD-L1 antibodies and explore the prognosis-relevant factors of advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically confirmed advanced solid tumors;
* Received anti-PD-1/PD-L1 antibody therapy.

Exclusion Criteria:

* No specific exclusion criteria in this real world study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced solid tumors who visited Department of Medical Oncology, Chinese PLA General Hospital from 2015 to 2019 and received anti-PD-1/PD-L1 antibody therapy
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-12-30 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 6 months
  PFS was defined as the length of time from the administration of the first-dose until disease progression or death from any cause before disease progression.

SECONDARY OUTCOMES:
Rate of adverse events (AEs)/ serious adverse events (SAEs) in patients with advanced solid tumors receiving anti-PD-1/PD-L1 antibody therapy. | up to 4 weeks after the last dose
  AEs/SAEs were evaluated using NCI-CTCAE v5.0
Objective Response Rate (ORR) | 6 months
  ORR was defined as the percentage of patients with complete response (CR) and partial response (PR) according to Response Evaluation Criteria in Solid Tumours (RECIST).
Disease Control Rate (DCR) | 6 months
  DCR was defined as the percentage of patients with complete response (CR), partial response (PR) and stable disease (SD) according to Response Evaluation Criteria in Solid Tumours (RECIST).
Overall survival (OS) | up to 12 months
  OS was defined as the length of time from the administration of the first-dose until death from any cause.

OTHER OUTCOMES:
Biomarkers | before the first dose
  Explore the correlation between curative effect and different biomarkers, such as EGFR mutation, KRAS mutation, TMB and MSI

CONTACTS AND LOCATIONS:
Overall Officials: Shunchang Jiao, PhD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No